CLINICAL TRIAL: NCT01906515
Title: Continuous and Noninvasive Hemoglobin Monitoring Reduces Red Blood Cell Transfusion During Neurosurgery: A Prospective Cohort Study
Brief Title: Impact of SpHb Monitoring on Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, wael awada, Assistant Lecturer Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: doctor19
Record Dates: First submitted 2013-07-13; First posted 2013-07-24 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Anemia
Keywords: Anemia; Blood transfusion; non invasive hemoglobin monitoring; patient safety
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Control Group received standard anesthesia care including intraoperative blood sampling when estimated blood loss was ≥15% of total blood volume and transfusion when hemoglobin was ≤10 g/dL.
- SpHb Group. (Experimental): Continuous non-invasive hemoglobin monitoring (SpHb monitoring) was provided to the anesthesiologist to influence administration of care
  Interventions: Device: Continuous non-invasive hemoglobin monitoring

INTERVENTIONS:
Device: Continuous non-invasive hemoglobin monitoring — Anesthesiologist is provided with real-time continuous non-invasive hemoglobin monitoring to influence care provided to patient
  Other Names: Masimo Radical-7 with SpHb
  Arms: SpHb Group.

SUMMARY:
Continuous and noninvasive hemoglobin (SpHb) monitoring provides clinicians with real-time trending of changes or lack of changes in hemoglobin, which has the potential to alter red blood cell (RBC) transfusion decision making. The objective of this study was to evaluate the impact of SpHb monitoring on RBC transfusions in high blood loss surgery. The investigators hypothesize that SpHb will improve blood transfusion practice in the for of change the number of blood unit per patient and improve the outcome regards the time to take decision of transfusion trigger.

DETAILED DESCRIPTION:
Eligible patients scheduled for neurosurgeries were enrolled into either a standard care group (Control Group) or an intervention group (SpHb Group). The Control Group received typical anesthesia care including estimated blood loss (EBL) assessment and intraoperative hemoglobin measurements from the central laboratory (Hb). Blood samples were taken when EBL was ≥15% of total blood volume. RBC transfusion was initiated if Hb was ≤10 g/dL and continued until the EBL was replaced and Hb >10g/dL was confirmed. The SpHb Group followed the same transfusion practice as the Control Group except the anesthesiologist was guided by the addition of SpHb monitoring with blood samples still taken pre- and post-transfusion. Additionally, the absolute and trend accuracy of SpHb compared to Hb was evaluated. Potential cost savings from reduced RBC utilization will be calculated if occured.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1,2 patients from 15 to 60 years old scheduled for neurosurgical procedure

Exclusion Criteria:

* Exclusion criteria included significant liver or renal disease, coagulopathy, pregnancy, anemia, and patients scheduled for procedures with excepted low blood loss.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wael N Awada, MD, Principal Investigator — Department of Anesthesia, ICU, and Pain Management, Cairo University, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for neurosurgery
Groups:
- SpHb Group.: In the SpHb Group, the anesthesiologist was guided by the addition of SpHb monitoring.
  Continuous non invasive hemoglobin monitoring arm
  continuous non invasive hemoglobin monitoring : Masimo radical pulse co oximetry
Period: Overall Study
Arm/Group | SpHb Group. | Control Group
Started | 45 | 61
Completed | 45 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SpHb Group. | Control Group | Total
Number analyzed (Participants) | 45 | 61 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 39 | 55 | 94
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 56
  Male | 20 | 30 | 50
Region of Enrollment [Number; unit: participants]
  Egypt | 45 | 61 | 106

OUTCOME MEASURES:

1. Secondary Outcome: SpHb Absolute and Trend Accuracy
Description: To assess absolute accuracy, or single point comparison, paired SpHb and Hb measurements were compared pre- and post- transfusion and bias and standard deviation were calculated. A Bland Altman graph with limits of agreement (1.96 x standard deviation, adjusted for the bias) was plotted to show agreement across the range of values. To assess trending, a regression plot of changes in Hb and corresponding changes in SpHb was plotted and a coefficient of determination (R2) was calculated
Time Frame: During surgery (an average of about 4 hours)
Reporting Status: Not Posted

2. Other Pre Specified Outcome: Potential Cost Savings
Description: Potential cost saving resulting from reduced RBC utilization was estimated using activity-based cost estimates established by Shander et al.(8) which determined from both U.S. and European hospitals the total cost of transfusing one RBC unit to be between $522 and $1,183 with a mean and standard deviation of $761 ± $294.
Time Frame: During surgery (an average of about 4 hours)
Reporting Status: Not Posted

3. Primary Outcome: RBC Transfusions Per Subject Receiving a Transfusion
Description: Determine whether using SpHb can affect the quantity of RBC transfused, per patient receiving a transfusion.
Time Frame: During surgery (an average of about 4 hours)
Population: We only included the participants who received a blood transfusion during the surgery for this analysis. Participants who did not receive a transfusion were excluded from this analysis.
Measure: Mean (95% Confidence Interval); unit: units
Arm/Group | SpHb Group. | Control Group
Number analyzed (Participants) | 19 | 30
units | 2.3 [1.6 to 3] | 3.9 [3.2 to 4.5]
Statistical Analysis 1: Comparison: SpHb Group. vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

4. Primary Outcome: The Effect of SpHb on Transfusion Timeline
Description: Length of time it takes to initiate a RBC transfusion after the need was first established.
Time Frame: During surgery (an average of about 4 hours)
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: minutes
Groups:
- SpHb Group.: In the SpHb Group, the anesthesiologist was guided by the addition of SpHb monitoring.
  Continuous non invasive hemoglobin monitoring arm.
  Continuous non invasive hemoglobin monitoring : Masimo radical pulse co oximetry
Arm/Group | SpHb Group. | Control Group
Number analyzed (Participants) | 19 | 30
minutes | 9.2 [8.4 to 10] | 50.2 [47.3 to 53]
Statistical Analysis 1: Comparison: SpHb Group. vs Control Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During surgery (an average of about 4 hours)
Arm/Group | SpHb Group. | Control Group
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/61
Other Adverse Events (participants affected / at risk) | 0/45 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes